CLINICAL TRIAL: NCT04373928
Title: A Single-centric, Prospective, Open, Interventional Clinical Trial, About Personalized Precision Diagnosis and Treatment of Pancreatic Cancer
Brief Title: Personalized Precision Diagnosis and Treatment of Pancreatic Cancer
Acronym: PPDTPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Attending surgeon at the Institute of Pancreatic surgery, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH-PP02
Record Dates: First submitted 2019-11-07; First posted 2020-05-05 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Cancer
Keywords: PDX,Mini-PDX,ctDNA,Conditional Reprogramming cells
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: According to randomized principles, patients with pancreatic cancer will be assigned to intervention group. Collecting the tumor tissue of intervention group and testing the best medicine by Mini PDX, which the person of intervention group receive the best medicine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug guided by Mini-PDX/PDX (Experimental): Procedure: The tumor tissue is used for drug sensitivity test by Mini-PDX, building PC PDX, and acquiring the genetic information by the second genetic sequence or RNA-sequence. PC patients will accept personalized treatment guided by the experimental results of mini-PDX and sequencing.
  Interventions: Procedure: Drug guided by Mini-PDX/PDX
- Drug according to guideline (No Intervention): The drugs (gemcitabine, Nab-paclitaxel, S-1) are used ccording to NCCN pancreatic cancer guideline。

INTERVENTIONS:
Procedure: Drug guided by Mini-PDX/PDX — Chemotherapeutic agents guided by Mini-PDX/PDX will be applied to PC patients and the efficiency will be studied.
  Other Names: Mini-PDX/PDX
  Arms: Drug guided by Mini-PDX/PDX

SUMMARY:
Pancreatic cancer (PC) is the 4th common cancer in the world and occupied the second place for digestive tumors, of which the incidence has also increased sharply in China. It harbors a particularly poor prognosis due to the late onset of symptoms and the advanced stage that the disease usually reaches before diagnosis. Therefore, searching more sensitive and accurate tumor markers has great value for application.

Circulating tumor cell (CTC) is a noninvasive index that could help diagnosis and monitor the load of tumor, having excellent prospect for clinical application. Early in the formation and growth of a primary tumor (breast, colon, lung, or prostate cancer, et al.), CTC are released into blood. The published studies on CTCs have focused on their prognostic significance, utility in real-time monitoring of therapies, resistance targets and understanding the process of metastasis. Our main purpose is to use the platform to identify correlations between CTC counts and PC progression.

Chemotherapy plays an important role in the postoperative treatment for PC. However, the efficiency of chemotherapeutic drugs for PC remains relatively limited. Patient-derived xenograft (PDX) preferably reproduce the clinical biological characteristics of PC, leading that we could deeply study the pathogenesis and metastasis of PC. Moreover, using PDX platform defines drug-resistant PC. From the present study, PDX and Mini-PDX platforms maintained architectural characteristics of the original PC specimen after continuous passaging, which could reflect the preclinical medicine study, better serving the clinical chemotherapy and improving the treatment efficiency.

Conditional reprogramming (CR) technique adds no virus or cell oncogene to the non-genetic operation, which will not change any gene phenotype during normal growth and continuous passage of the cells in vitro. After a small sample of PC patient is obtained by CR, the project could enlarge the tumor samples from micro-biopsy tissue samples, and provide a basis for the follow-up of tumor drug susceptibility testing. This experiment also uses ctDNA (circulation tomor DNA)technology to detect the genetic information of PC, through which it is expected to improve personalized precision diagnosis and treatment of PC and help to establish a complete database of individual PC PDX. It provides ideal research materials and platform for basic development and translational medicine research of oncology.

DETAILED DESCRIPTION:
Tumor cells are released from the primary tumor and/or metastatic sites into blood. Circulating tumor cells (CTC), as a part of liquid biopsy, is acted as a new method to diagnose cancer. Many studies indicated that CTC counts had a correlation with breast, colon, lung, or prostate cancer development. When individual cells or clusters of cancer cells acquire ability to separate and move away from the primary tumor, migrate through the surrounding tissue, and enter the lymphatic system and/or blood circulation, the metastatic trait of the given tumor become obvious [1-3]. Tumor cells that escape from their primary microenvironment need to avoid anoikis and might be challenged by the host's immunologic defense. Finally, CTC is like a seed that transfer to other organs, contributing to metastasis and recurrence. These CTC could be enriched and detected via different technologies that take advantage of their physical and biologic properties. This study collected CTC by iset platform which checks CTC (pre-operative\postoperative\pre-treatment\during treatment) and observed the association between CTC counts and PC development [4].

Patient-derived xenograft (PDX) was demonstrated to consistently retained tumor morphology and genetic phenotype. Different from traditional cell line xenotransplantation model and genetically engineered mouse model, pancreatic adenocarcinoma specimens were engrafted to immuno-deficient mice. Above all, PDX could keep special functional gene structure and biomarkers in personal case, closer to the individual clinical biological characteristics and providing better prediction effect for drug screening and observation for treatment efficiency.

As some researches discovered, the effective of contrasting drug sensitivity test with clinical drug response is >90% [5]. Now, we build the PDX of PC, checking the genetic information by the second genetic sequence or RNA-sequence. If PDX has similar genetic information to the primary tumor, we will do drug sensitivity test. PC PDX model, whereby we have demonstrated that the early PDX was morphologically similar to the original cancer and retained both inter-patient and intra-patient heterogeneity of the tumor, could provide reference model for personalized treatment of PC.

Above all, the most obvious advantage of PDX is the similarity to primary tumor, so we could check the sensitivity of the same drug. But building PDX will take about 3-4months (including building the model and drug sensitivity test). As a result, we need clinical precision therapeutic plan applying to the developed pancreatic cancer patients. Miniature Patient Derived Xenograft (Mini-PDX), from Shanghai LIDE(lide) Biotech CO(company), was carried out with the OncoVeeTM-Mini PDX product of LIDE Biotech, and followed the instruction from the manufacturer. Tumor samples were harvested, and washed with HBSS(Hank's balanced salt solution) to remove non-tumor tissue and necrotic tumor tissue in biosafety cabinet. After the tumor samples were cut into small fragments, they were incubated with collagenase solution at 37℃ for 1-2 hours. Then we collected the cells followed by removing the blood cells and fibroblast cells and the cell suspension was transferred to the HBSS washed capsules. For subcutaneous (s.c.) implantation, a small skin incision was made and the capsule was inserted through the subcutaneous tissue. Generally, each mouse received 4 capsules and drug administration was carried out for 7 days. The anti-tumor activity was evaluated through the CTG (cell viability) assay.

The combination of irradiated fibroblast feeder cells and Rho kinase inhibitor, Y-27632, conditionally induced an indefinite proliferative state in primary mammalian epithelial cells. These conditionally reprogrammed cells (CRCs) were karyotype-stable and nontumorigenic. Because self-renewal was a recognized property of stem cells, we investigated whether Y-27632 and feeder cells induced a stem-like phenotype. We found that CRCs shared characteristics of adult stem cells and exhibited up-regulated expression of α6 and β1 integrins, ΔNp63α, CD44, and telomerase reverse transcriptase, as well as decreased Notch signaling and an increased level of nuclear β-catenin. The induction of CRCs was rapid (occurs within 2 d) and resulted from reprogramming of the entire cell population rather than the selection of a minor subpopulation. CRCs did not overexpress the transcription factor sets characteristic of embryonic or induced pluripotent stem cells (e.g., Sox2, Oct4, Nanog, or Klf4). The induction of CRCs was also reversible, and removal of Y-27632 and feeders allowed the cells to differentiate normally. CRCs was called on the news human precision protocol. In the pancreatic cancer precision study, patients with inoperable or developed who acquired a little tissue could not build PDX and lost the chance of PDX treatment. Hence, we used the CRCs platform to grew tumor stem cell in vitro, when having adequate cells, we could do Mini-PDX or PDX drug assay[6].

In summary, as different stages of PC patients could not acquire precision personalized in clinical treatment at present, this study by CTC\PDX\Mini-PDX\CRs\RNA-SEQ\NGS (Next generation sequencing)platforms were predicted to provide precision diagnosis and treatment for different stages of PC patients. Meanwhile, we could build tumor information biobank, which provided ideal research materials and platforms for oncology basic research and translational medicine research.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing radical resection of pancreatic cancer;
* No serious underlying disease;
* No preoperative chemotherapy;
* The diagnosis of pancreatic cancer;
* No significant heart, lung or renal function;
* No HIV or syphilis infection;
* All patients should sign the informed consent.

Exclusion Criteria:

* Preoperative general condition was poor, and it was estimated that the operation and postoperative chemotherapy and targeted therapy could not be tolerated;
* Patients with unstable angina pectoris, symptomatic congestive heart failure, severe arrhythmia, cardiac infarction in the past 6 months, and prolonged QT interval (>450ms).
* Patients with other malignancies in the last 5 years.
* Patients are not subject to follow-up or other clinical trials.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | up to 24 months
  Observing and comparing OS (overall survival time) between two groups.

SECONDARY OUTCOMES:
DFS | up to 24 months
  Observing and comparing DFS (disease free survival time) between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Gang, M.D., Study Chair — Department of general surgery, Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Result] Cohen SJ, Punt CJ, Iannotti N, Saidman BH, Sabbath KD, Gabrail NY, Picus J, Morse M, Mitchell E, Miller MC, Doyle GV, Tissing H, Terstappen LW, Meropol NJ. Relationship of circulating tumor cells to tumor response, progression-free survival, and overall survival in patients with metastatic colorectal cancer. J Clin Oncol. 2008 Jul 1;26(19):3213-21. doi: 10.1200/JCO.2007.15.8923. PMID 18591556
- [Result] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Result] Fiebig HH, Maier A, Burger AM. Clonogenic assay with established human tumour xenografts: correlation of in vitro to in vivo activity as a basis for anticancer drug discovery. Eur J Cancer. 2004 Apr;40(6):802-20. doi: 10.1016/j.ejca.2004.01.009. PMID 15120036
- [Result] Suprynowicz FA, Upadhyay G, Krawczyk E, Kramer SC, Hebert JD, Liu X, Yuan H, Cheluvaraju C, Clapp PW, Boucher RC Jr, Kamonjoh CM, Randell SH, Schlegel R. Conditionally reprogrammed cells represent a stem-like state of adult epithelial cells. Proc Natl Acad Sci U S A. 2012 Dec 4;109(49):20035-40. doi: 10.1073/pnas.1213241109. Epub 2012 Nov 19. PMID 23169653